CLINICAL TRIAL: NCT07190729
Title: Monocentric Randomised Controlled Trial to Assess Whether Virtual Reality Reduces the Use of Hypnotic Agents During IVF/ICSI Oocyte Retrieval
Acronym: REVAHPOVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A00311-42
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Medically Assisted Procreation (MAP); Oocyte Retrieval
Keywords: Virtual reality; Propofol sedation

STUDY DESIGN:
Intervention Model Description: Control group: standard propofol sedation procedure Experimental group: standard propofol sedation procedure + mask -RV Deepsen™
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Control group: the participants will receive standard propofol sedation procedure
  Interventions: Other: Propofol sedation
- Experimental arm (Experimental): Experimental group: the participants will receive standard propofol sedation procedure and the mask -RV Deepsen™
  Interventions: Device: Propofol sedation + Audiovisual distraction

INTERVENTIONS:
Device: Propofol sedation + Audiovisual distraction — The participants will receive standard propofol sedation procedure and the mask -RV Deepsen™
  Arms: Experimental arm
Other: Propofol sedation — The participants will receive standard propofol sedation procedure
  Arms: Control arm

SUMMARY:
Over the last few years, audiovisual distraction devices using animation, films and 3D immersion have been developed, with the aim to provide patients with a relaxing experience that disconnects them from the operating environment while still allowing them to interact with the surgeon. These devices make it easier for surgeons to perform short procedures and improve patients' experiences.

Virtual distraction techniques have been evaluated in several areas, particularly in managing preoperative pain and anxiety in adults.

However, to date, no study comparing different techniques for focusing attention and the anaesthetic management of oocyte punctures has been published. Our study will evaluate if using the Deepsen™ mask device to focus attention in a virtual reality environment is more effective than the usual verbal reassurance technique at reducing anxiety levels and sedation requirements during oocyte punctures, while improving comfort and enabling faster walking.

DETAILED DESCRIPTION:
Over the last few years, audiovisual distraction devices using animation, films and 3D immersion have been developed. These devices aim to provide patients with a relaxing experience that disconnects them from the operating environment while still allowing them to interact with the surgeon. These devices make it easier for surgeons to perform short procedures and improve patients' experiences.

Virtual distraction techniques have been evaluated in several areas, particularly in managing preoperative pain and anxiety in adults.

However, no study comparing different techniques for focusing attention and the anaesthetic management of oocyte punctures has been published to date. This study hypothesises that using the Deepsen™ mask device to focus attention in a virtual reality environment is more effective than the usual verbal reassurance technique at reducing anxiety levels and sedation requirements during oocyte punctures, while improving comfort and enabling faster walking.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 and under 43 years of age.
* Requiring propofol sedation for oocyte puncture.
* Who can be contacted directly by telephone the day after the procedure.
* Have given their consent to participate in accordance with the regulations.
* Benfeting of a social security scheme or entitled persons (excluding AME).

Exclusion Criteria:

* Active endometriosis.
* Presence of at least one anatomically high ovary which is difficult to puncture.
* Inability to understand the information provided.
* Under guardianship, curatorship or legal protection.
* Under psychiatric care.
* Admitted to a health or social establishment for purposes other than this research.
* Under constraint or deprived of liberty by judicial or administrative decision.
* Impaired communication or neuropsychological disorders.
* Ongoing corneal or conjunctival pathologies.
* Claustrophobia.
* Nausea in the mountains or at sea.
* Use of an anxiolytic or sleeping pill in the 12 hours prior to randomisation.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The Cp50 value of propofol in each group. | Day 0
  The Cp50 is defined as the median of the target concentration at which 50% of participants showed movement during the oocyte puncture procedure. Any difference between the two groups will be determined using Dixon's up and down technique
The number and proportion of participants not requiring sedation | Day 0

SECONDARY OUTCOMES:
Effect on procedural anxiety | Day 0
  The participant's anxiety was measured prior to the study. It was assessed using the STAI questionnaire in order to define the general state of anxiety (STRAI) and the level of immediate anxiety in relation to the examination (STATE). This is a two-part questionnaire with around thirty questions in each section, for which a single response is used to describe the intensity of the relationship: very often, often, rarely, never. An anxiety VAS will be requested at the time of the WHO checklist, together with the intensity of any pain. These questions will be asked again in the intensive care unit when the patient is put in the standing position.
Tolerating audiovisual distraction | 48 hours
  Tolerance of the device and the audiovisual distraction session is defined by the occurrence of undesirable effects (dizziness, nausea, headaches). This is done using a 4-level scale for each item (none, mild, moderate, severe).
Pain on injection of propofol | Day 0
  The intensity of pain on propofol injection was assessed using a three-point behavioural scale for facial expression (0: none, 1: frown, or 2: grimace), verbal response (0: none, 1: groan, or 2: clear expression of pain) and attempt to withdraw the arm (0: none, 1: medium, or 2: strong). The discomfort scale is the sum of these three clinical parameters and therefore ranges from 0 to 6.
Complications observed during anaesthesia | Day 0
  Any complications linked to anaesthesia from induction to recovery are collected:
  * Number of events with arterial oxygen desaturation below 92%,
  * Number of episodes with a ventilatory frequency of less than 10 cycles/min,
  * Occurrence of bronchospasm.
The time required to walk | Day 0
  Time to street readiness will be assessed using the CHUNG
Acceptance of audiovisual distraction by anaesthetists, gynaecologists and other healthcare professionals | Day 0
  Acceptance of audiovisual distraction by anaesthetists, gynaecologists and nursers will be assessed using a 4-level scale (very satisfied, satisfied, partially satisfied, not satisfied) and by collecting reasons for not being satisfied (partially satisfied, not satisfied) (short open answers).
Participant satisfaction with the procedure | Day 0
  Participant satisfaction is assessed on leaving the post-interventional monitoring room using a 4-level scale (very satisfied, satisfied, partially satisfied, not satisfied), with a free text provided in addition. Any interruption of the audiovisual distraction session at the participant's request will be noted. Satisfaction with the procedure may also be obtained from healthcare professionals.
Resumption of activities of daily living | Day 1
  Resumption of activities of daily living was assessed during the next day's telephone call using a subjective numerical rating scale ranging from 0 (bedridden) to 10 (full recovery).
Recovery room discharge time | Day 0
  Post-intervention monitoring room discharge time is defined as the time between the end of the operation and the achievement of an ALDRETE score of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No